CLINICAL TRIAL: NCT04051398
Title: Effects of Transcutaneous Nerve Electrostimulation (TENS) of Acupuncture Points on Pulmonary Function and Dyspnea Symptoms in Patients With Pulmonary Nodules Treated at a Referral Service: A Randomized Single Blind Study
Brief Title: Effects of Transcutaneous Nerve Electrostimulation (TENS) of Acupuncture Points on Pulmonary Function and Dyspnea Symptoms in Patients With Pulmonary Nodules
Acronym: LUNG TENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Santa Marcelina (Other)
Responsible Party: Principal Investigator, Igor Renato Louro Bruno de Abreu, Medical Staff of Thoracic Surgery Department of Santa Marcelina Hospital, Hospital Santa Marcelina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Santa Marcelina Hospital
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Lung Diseases; Dyspnea; Acupuncture
Keywords: Acupuncture; Lung
MeSH Terms: conditions — Lung Diseases; Dyspnea | interventions — Transcutaneous Electric Nerve Stimulation; Acupuncture Points

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: . To minimize the impact of non-blinding investigators, will be designated a specific investigator who will be responsible for randomizing participants at the time of TENS application and performing the intervention do not allowing the investigators responsible for data collection know whether the patient will be BI or BC. After data collection, the same investigator will segregate the information from BC and BI keeping the subgroups identification in secret do not allowing the investigator who will perform the statistical analysis know what are the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (BI) (Experimental): The BI participants will initially undergo simple spirometry and a 6-minute walk test and Borg scale application upon admission to the thoracic surgery department. Immediately after the exams, they will undergo a TENS application session over the acupuncture points: Feishu, Zhongfu, Taiyuan and Dingchuan using a frequency of 200Hz and a pulse time of 80 seconds of sufficient intensity to cause a slight sensation of local numbness without muscle fasciculations. The TENS application time will be 30 minutes. Immediately after the TENS application, the participants will be submitted to a new spirometry, a new 6-minute walk test and again to the Borg scale.
  Interventions: Other: transcutaneous nerve electrostimulation (TENS) of acupuncture points
- Control Arm (BC) (Placebo Comparator): The BC participants will undergo the same steps as BI, however when applying TENS to these participants investigators will place the electrodes over the points without turning on the device in order to obtain the effect of a placebo.
  Interventions: Other: transcutaneous nerve electrostimulation (TENS) of acupuncture points

INTERVENTIONS:
Other: transcutaneous nerve electrostimulation (TENS) of acupuncture points — TENS application session over the acupuncture points: Feishu, Zhongfu, Taiyuan and Dingchuan using a frequency of 200Hz and a pulse time of 80 seconds of sufficient intensity to cause a slight sensation of local numbness without muscle fasciculations. The TENS application time will be 30 minutes.
  Other Names: TENS Acupuncture

SUMMARY:
The ancient use of acupuncture as a treatment modality of traditional Chinese medicine has also been proven effective in Western medicine. The use of this treatment tool for pain control is already proven in the literature and today is considered an important adjuvant for this purpose. However, the ancient texts of acupuncture also report the use of certain points to tonify organs functions, despite of pain control. According to these texts there are some points that allow the treatment of lung diseases improving respiratory function.

In order to investigate the effects of stimulation of such points using electric field application, the effect of these procedure on pulmonary function and the impact of this practice on dyspnea symptoms, the investigators will conduct a randomized study with 60 patients (1: 1 randomization) distributed in 2 arms (intervention arm-BI and control arm-BC). Transcutaneous neural stimulation of acupuncture points of the BI patients will be performed. For the BC arm the investigators will place the electrodes over the points without turn on the device to produce a placebo effect. Pulmonary function test, Borg scale application and 6 min walk test will be performed before and after the intervention in each group for subsequent data comparison.

DETAILED DESCRIPTION:
Introduction:

The use of acupuncture for pain management is well defined and fully established. The stimulation of acupuncture points using needles, electrical stimuli, thermal or laser stimuli produce local effects at the point (nociceptor stimulation and release of inflammatory mediators) that generate systemic effects (serotonin release and endorphins in the Central Nervous System). leading to the state of body relaxation, well-being, changes in heart rate, blood pressure and analgesia.

However, acupuncture can trigger other effects beyond pain control. In ancient texts dealing with the subject there are descriptions of points capable of promoting improvement of specific organic functions such as pulmonary function. 2 This effect is due to changes generated by the action of acupuncture on the autonomic nervous system promoting bronchodilation and decreased mucus production. Some studies of effects of acupuncture in patients with chronic obstructive pulmonary disease have shown promising results related to improved lung function and reduced symptoms.

Transcutaneous nerve electrostimulation (TENS) can be used to stimulate acupuncture points as an alternative to needles. This modality of stimulation prevents the occurrence of serious complications such as pneumothorax secondary to needle application to thoracic points. This practice turns the procedure safer allowing any trainned healthcare professional to do it.

Goals:

1. Evaluate the immediate effects of this procedure on pulmonary function.
2. Evaluate the effects of TENS on dyspnea symptoms.

Materials and methods:

Will be recruited 60 participants over the age of 18 years, smokers and patients with pulmonary nodules attended at Santa Marcelina Hospital. Patients with pacemakers, patients unable to read, understand and sign the informed consent form, with mobility restrictions, chest pain and patients who have previously used TENS will be excluded from this study.

Participants will be randomized in a 1/1 ratio to form 2 arms: intervention arm (BI) and control arm (BC).

The BI participants will initially undergo simple spirometry and a 6-minute walk test and Borg scale application (this texts are detailed at "Tests Description" item at the end of this manuscript) upon admission to the thoracic surgery department. Immediately after the exams, they will undergo to a TENS application session over the acupuncture points: Feishu, Zhongfu, Taiyuan and Dingchuan using a frequency of 200Hz and a pulse time of 80 seconds of sufficient intensity to cause a slight sensation of local numbness without muscle fasciculations. The TENS application time will be 30 minutes. Immediately after the TENS application, the participants will be submitted to a new spirometry, a new 6-minute walk test and again to the Borg scale evaluation.

The BC participants will undergo to the same steps as BI, however when applying TENS to these participants the investigators will place the electrodes over the points without turning on the device in order to obtain the effect of a placebo. To minimize the impact of non-blinding investigators, will be designated a specific investigator who will be responsible for randomizing participants at the time of TENS application and performing the intervention do not allowing the investigators responsible for data collection know whether the patient will be BI or BC. After data collection, the same investigator will segregate the information from BC and BI keeping the subgroups identification in secret do not allowing the investigator who will perform the statistical analysis know what are the groups. Once the data analysis is ready, the investigator responsible for randomization will tell the other investigators which subgroup corresponds to each arm.

Tests Description:

# 6-minute Walk Test (6 MWT):

In 2002, the American Thoracic Society (ATS) published guidelines on how to perform the 6 MWT. This guideline stressed the need for a standardized protocol to perform the 6 MWT to minimize variation in results.

Although the 6 MWT is very safe, emergency equipment should be at hand. The test should be conducted by personnel qualified to use this equipment. Physicians are not required to be present in most situations, but should be readily available. The physician ordering the test may decide if a physician should supervise the test.

According to ATS guidelines, a 30 meters distance course is recommended. Turnaround points should be identified. Three-meter interval measurements are marked with colored tape on the floor. Shorter corridor lengths may increase the 6 MWD due to more frequent turns involved.

Required equipment

1. Stop watch or timer
2. Two small cones to mark the lap boundaries
3. Measurement scale for floor measurement
4. Mechanical lap counter
5. Resuscitation equipment

The 6 MWT is performed on a walking track in hospital facility. The track has been marked at 3-m intervals so that accurate measurement of the walking distance can be performed. Chairs are available at 30-m intervals in case the patients become so symptomatic that have to stop and sit.

Patient preparation

1. Comfortable clothing should be worn
2. Environment temperature should be ambient
3. Shoes should be comfortable and any walking aids that the patient ordinarily uses should be used
4. Light meals are acceptable before morning and afternoon tests

Technique

1. Don't perform a warm up before the test.
2. The patient should rest comfortably for 10 minutes prior to the test. During this time blood pressure and heart rate should be measured and potential contraindications assessed.
3. Pulse oximetry is optional. If it is used, it should be ensured that readings are stable prior to starting the 6 MWT, and signal is optimized.
4. Before the test starts, the patient should stand up and rate for dyspnea and fatigue. The Borg scale may be used for this.
5. Set the lap counter to zero and timer to 6 minutes. Assemble all necessary equipment and move to starting point.
6. The supervisor may walk a lap to demonstrate performance of the test to the patient. During the test the supervisor should never walk with or in front of the patient as the patient may try to match the supervisor's pace. The supervisor may walk behind the patient to support the patient in case of staggering or to prevent falling. The patient is allowed to rest during the test if gets fatigued.
7. Use standardized phrases and an even tone for encouragement at completion of each minute of the test. For an example of a standardized script, the reader is referred to the 2002 ATS guidelines. Some examples are "keep up the good work" or "you are doing fine".
8. Resting during the test is allowed, but don't stop the clock. If the patient cannot go any further, the test should be stopped and distance covered recorded.
9. Stop the test if patient develops chest pain, intolerable dyspnea, staggering, diaphoresis, intolerable cramps, and/or ashen appearance. Test supervisors should be trainned to provide appropriate care at this point.
10. At the conclusion of the test, ask the patient to rate his/her dyspnea and fatigue levels. Record the reason for stopping the test.

Additional details about technique

1. If the patient is on supplemental oxygen, use the same oxygen level that normally uses with exercise.
2. The 2002 ATS guidelines do not recommend routine measurement of pulse oximetry during the test. In untreated patients with pulmonary hypertension, oxygen desaturation >10% during 6 MWT has been associated with mortality. With the widespread availability of light-weight portable oximeters, monitoring of oxygen saturation during walking can be reliably performed.
3. Quality control and standardization are important to reduce variability in measurement. Persons supervising the test should be trained using a standard protocol, and should conduct supervised 6 MWTs before patients are able to perform them independently. A practice test generally should not be needed. If a practice test is done, there should be a wait time of about an hour between the two tests, and the longer 6 MWD should be reported.

   * Borg scale measure:

The scale allows individuals to subjectively rate their level of exertion during exercise or exercise testing.

It is a gradual scale that varies from zero (no fatigue symptoms) to ten (maximum fatigue like the sensation of the hardest race that the participant have ever did)

Patients with higher values on Borg scale evaluation are considered worse.

see the link of Borg scale at the references.

ELIGIBILITY:
Inclusion Criteria:

* smokers
* patients with pulmonary nodules attended at Santa Marcelina Hospital.

Exclusion Criteria:

* Patients with pacemakers
* patients unable to read, understand and sign the informed consent form
* patients with mobility restrictions
* patients with chest pain
* patients who have previously used TENS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the immediate effects of this procedure on forced expiratory volume in one second (FEV1). | 45 minutes after the beginning of intervention of each participant.
  To evaluate this outcome the investigators will access the forced expiratory volume in one second (FEV1) values from the spirometry prior to intervention and post intervention spirometry to compare if there are diferences in these values after the TENS application or placebo according to the subgroup of each participant
Evaluate the immediate effects of this procedure on forced vital capacity (FVC). | 45 minutes after the beginning of intervention of each participant.
  To evaluate this outcome the investigators will access the forced vital capacity (FVC) values from the spirometry prior to intervention and post intervention spirometry to compare if there are diferences in these values after the TENS application or placebo according to the subgroup of each participant
Evaluate the immediate effects of this procedure on VEF1/FVC ratio. | 45 minutes after the beginning of intervention of each participant.
  To evaluate this outcome the investigators will access the VEF1/FVC ratio values from the spirometry prior to intervention and post intervention spirometry to compare if there are diferences in these values after the TENS application or placebo according to the subgroup of each participant
Evaluate the immediate effects of this procedure on 6 - minute Walk Test. | 45 minutes after the beginning of intervention of each participant.
  To evaluate this outcome the investigators will access the 6 minutes Walk Test distance values prior to intervention and post intervention to compare if there are diferences in these values after the TENS application or placebo according to the subgroup of each participant
Evaluate the effects of TENS on dyspnea symptoms. | 45 minutes after the beginning of intervention of each participant.
  The investigators will compare the Borg scale measures prior and after the intervention to access if the were changes in dyspnea symptoms for each participant from each arm.

SECONDARY OUTCOMES:
Evaluate the effects of TENS on blood oxygen saturation. | 45 minutes after the beginning of intervention of each participant.
  The investigators will compare the blood oxygen saturation using the pulse oximetry measures prior and after the intervention to access if the were changes in dyspnea symptoms for each participant from each arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Ambulatório de Nódulos e Massas Pulmonares H Santa Marcelina, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu L, Chen S, Zeng D, Li H, Shi C, Zhang L. Cerebral activation effects of acupuncture at Yanglinquan(GB34) point acquired using resting-state fMRI. Comput Med Imaging Graph. 2018 Jul;67:55-58. doi: 10.1016/j.compmedimag.2018.04.004. Epub 2018 Apr 21. PMID 29800886
- [Background] Xing X, Wang Y, Cui L, Liang Y. [Professor GAO Yuchun's understandings of "treating spirit" and "acupuncture reinforcing and reducing" in Inner Canon of Yellow Emperor and clinical experience]. Zhongguo Zhen Jiu. 2017 Feb 12;37(2):195-198. doi: 10.13703/j.0255-2930.2017.02.026. Chinese. PMID 29231486
- [Result] Suzuki M, Muro S, Ando Y, Omori T, Shiota T, Endo K, Sato S, Aihara K, Matsumoto M, Suzuki S, Itotani R, Ishitoko M, Hara Y, Takemura M, Ueda T, Kagioka H, Hirabayashi M, Fukui M, Mishima M. A randomized, placebo-controlled trial of acupuncture in patients with chronic obstructive pulmonary disease (COPD): the COPD-acupuncture trial (CAT). Arch Intern Med. 2012 Jun 11;172(11):878-86. doi: 10.1001/archinternmed.2012.1233. PMID 22905352
- [Result] Mehani SHM. Immunomodulatory effects of two different physical therapy modalities in patients with chronic obstructive pulmonary disease. J Phys Ther Sci. 2017 Sep;29(9):1527-1533. doi: 10.1589/jpts.29.1527. Epub 2017 Sep 15. PMID 28931981
- [Result] Johnson M. Transcutaneous Electrical Nerve Stimulation: Mechanisms, Clinical Application and Evidence. Rev Pain. 2007 Aug;1(1):7-11. doi: 10.1177/204946370700100103. PMID 26526976
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- See also: Borg Scale — https://doi.org/10.1378/chest.107.6.1590